CLINICAL TRIAL: NCT02878720
Title: Combining Non-Invasive Vagus Nerve Stimulation and Robotic Training in Upper Limb-Impaired Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Collaborators: Biomedical Robotics and Biomicrosystems, Campus Bio-Medico University (Unknown); Physical and Rehabilitation Medicine, Campus Bio-Medico University (Unknown)
Responsible Party: Principal Investigator, Di Lazzaro Vincenzo, Full Professor of Neurology, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VagusStroke
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: ischemic stroke; hemorrhagic chronic; non-invasive vagus nerve stimulation; robot-assisted rehabilitation
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic therapy and real tVNS (Experimental): This group receives REAL vagus nerve stimulation during robotic rehabilitation.
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Robotic therapy and sham tVNS (Active Comparator): This group receives SHAM VNS during robotic rehabilitation. Sham VNS is not effective. Both groups receive the same amount of robotic rehabilitation.
  Interventions: Device: Transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — The stimulation of the auricular branch of the vagus nerve will be performed through an electric stimulator and two Ag-AgCl electrodes placed in the left external acoustic meatus at the inner side of the tragus. For sham stimulation, electrodes will be attached to the left ear lobe. tVNS will be delivered as trains lasting 30 s and composed by 600 pulses (intra-train pulse frequency = 20 Hz; pulse duration = 0.3 ms) repeated every 5 min for 60 min. The intensity of stimulation will individually adjusted to a level ranging above the detection threshold and below the pain threshold. In this range, when possible, the investigators will chose an intensity of 8 mA.
  Each day, for 10 consecutive working days, each patient will receive a session of robotic therapy during the real or sham tVNS stimulation

SUMMARY:
Previous studies suggested that both robot-assisted rehabilitation and non-invasive vagus nerve stimulation can improve upper limb function in chronic stroke patients. Aim of present study is to explore whether the combination of these two approaches might enhance their positive effects on motor recovery. Safety and efficacy of this combination will be assessed within a proof-of-principle, double-blinded, randomized, sham-controlled trial. Transcutaneous vagus nerve stimulation (tVNS) will be delivered at left ear, in order to improve the response to the following robot-assisted therapy. Patients with both ischemic and hemorrhagic chronic stroke will be randomized to robot-assisted therapy associated with real or sham tVNS, delivered for 10 working days. Change in Fugl-Meyer has been chosen as primary outcome, while changes in several quantitative indicators of motor performance extracted by the robot as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* first-ever ischemic or hemorrhagic stroke at least 1 year earlier
* hand function impairment
* ability to give informed consent and comprehend instructions

Exclusion Criteria:

* previous surgical intervention on vagus nerve
* low hearth rate (< 60 bpm)
* cognitive impairment or any substantial decrease in alertness, language reception, or attention that might interfere with understanding instructions for motor testing
* apraxia
* excessive pain in any joint of the paretic extremity
* advanced liver, kidney, cardiac or pulmonary disease
* history of significant alcohol or drug abuse
* depression or use of neuropsychotropic drugs such as antidepressants or benzodiazepines
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Score | immediately, one months and three months after the intervention

SECONDARY OUTCOMES:
Change in kinematic data (Motion Accuracy) measured by the robot | immediately, one months and three months after the intervention
Change in kinematic data (Motion Direction) measured by the robot | immediately, one months and three months after the intervention
Change in kinematic data (Smoothness) measured by the robot | immediately, one months and three months after the intervention
Change in kinematic data (Speed) measured by the robot | immediately, one months and three months after the intervention
Change in kinematic data (Movement Duration) measured by the robot | immediately, one months and three months after the intervention
Change in kinematic data (Efficiency) measured by the robot | immediately, one months and three months after the intervention
Incidence of adverse events that are related to treatment | intervention period of 10 consecutive working days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Neurology, Campus Biomedico University, Rome, Italy

IPD SHARING:
Plan to Share IPD: No